CLINICAL TRIAL: NCT06856499
Title: Phase I Evaluation of Combination CLK/DYRK (Cirtuvivint) Inhibition With PARP Inhibition (Olaparib) in BRCA/HRD Platinum Resistant Ovarian Cancer
Brief Title: Cirtuvivint/Olaparib in Breast Cancer Susceptibility Gene/Homologous Recombination Deficiency Platinum Resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-1749.cc; R01CA288651-01 (NIH); NCI-2024-09126 (Other: CTRP)
Record Dates: First submitted 2025-01-13; First posted 2025-03-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Endometrioid Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Regimen 1 (Experimental): Patients on Dose Regimen 1 will take 300mg PO BID olaparib in combination with 80mg PO cirtuvivint for 5 days on and 2 days off.
  Interventions: Drug: Cirtuvivint; Drug: Olaparib
- Dose Regimen 2 (Experimental): Patients on Dose Regimen 2 will take 300 mg PO BID olaparib in combination with 120 mg PO cirtuvivint for 2 days on and 5 days off
  Interventions: Drug: Cirtuvivint; Drug: Olaparib

INTERVENTIONS:
Drug: Cirtuvivint — Cirtuvivint (SM08502) is a first in class pan CDC-like kinase (CLK) and dual specificity tyrosine kinase (DYRK) inhibitor with suspected multiple anti-tumor mechanisms of action, including Wnt inhibition.
Drug: Olaparib — NCI Definition - A small molecule inhibitor of the nuclear enzyme poly(ADP-ribose) polymerase (PARP) with potential chemosensitizing, radiosensitizing, and antineoplastic activities. Olaparib selectively binds to and inhibits PARP, inhibiting PARP-mediated repair of single strand DNA breaks; PARP inhibition may enhance the cytotoxicity of DNA-damaging agents and may reverse tumor cell chemoresistance and radioresistance. PARP catalyzes post-translational ADP-ribosylation of nuclear proteins and can be activated by single-stranded DNA breaks.
  Other Names: Lynparza

SUMMARY:
The purpose of this study is to learn about the safety and tolerability of Cirtuvivint in combination with Olaparib in platinum resistant ovarian cancer. The study also aims to determine the recommended dose of the combination therapy.

If a participant is a good fit for the study, and they enroll in the study, they will:

* Visit the clinic often at the beginning of the study for physical exams, blood draws, vital signs, and other study and routine care procedures. After the first two months participants will visit the clinic every 28 days.
* Take the study medications, Cirtuvivint and Olaparib. Participants will take Olaparib every day. Participants will either take Cirtuvivint 5 days per week or 2 days per week.

DETAILED DESCRIPTION:
This trial is a non-comparative phase I combination trial with the goal of determining the safety and RP2D of cirtuvivint when given orally daily (5 days on 2 days off) combined with olaparib given orally BID (continuously) for 28 day cycles, and of cirtuvivint when given orally daily (2 days on 5 days off) combined with olaparib given orally BID (continuously) for 28 day cycles. Patients will enter the two cohorts in alternating fashion by time of enrollment. The patient population will be women with platinum resistant high grade serous or endometrioid epithelial ovarian cancer who are germline or somatic BRCA/HRD positive. Due to potential survival detriment of late line PARP inhibition, patients will be limited to no more than 3 prior lines of therapy. Olaparib will be dosed at the standard recommended dose of 300mg BID and adjusted appropriately for known adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Woman aged ≥18 years of age
4. Patients must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 1 or 2
5. Patients must have a confirmed diagnosis of high-grade serous or endometrioid epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
6. Patients must have platinum-resistant disease defined as radiographic progression less than 6 months from last dose of most recent platinum therapy
7. Patients must have measurable disease by defined RECIST 1.1 criteria
8. Prior anticancer therapy:

   * Patients must have received at least one prior platinum-based chemotherapy regimen
   * Patients may not have received more than 3 prior lines of systemic therapy
   * Neoadjuvant +/- adjuvant therapies are considered 1 line of therapy
   * Maintenance therapy (eg, Bevacizumab, PARP inhibitors) will be considered part of preceding line of therapy (ie, not counted independently)
   * Therapy changed due to toxicity in the absence of progression will be considered part of the same line (ie, not counted independently)
   * Hormonal therapy will be counted as a separate line of therapy unless it was given as maintenance
   * Prior radiation is allowed and is not considered a line of treatment
9. Patients must have had testing for BRCA mutation (tumor or germline) and tumor HRD testing, and have been positive for one and/or the other.
10. Patients must have received a prior PARP inhibitor as either treatment or maintenance therapy
11. Patients must have adequate hematologic, liver, and kidney function as defined as:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/µL)
    * Platelet count ≥ 100 x 109/L (100,000 µL)
    * Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
    * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
    * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test
    * Aspartate aminotransferase (AST)(Serum Glutamic Oxaloacetic Transaminase (SGOT)) and alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x ULN unless liver metastases are present in which case they must be ≤ 5x ULN
    * Serum bilirubin ≤ 1.5 x ULN (patients with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0 x ULN)
    * Serum albumin ≥ 2 g/dL
12. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
13. Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible.

Exclusion Criteria:

1. Patients with clear cell, mucinous, sarcomatous, low grade/borderline, germ cell, or sex-cord stromal type ovarian tumor
2. Patients with platinum refractory disease as defined by those who have progressed during or within 4 weeks of receiving platinum-based therapy
3. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
4. Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome/acute myeloid leukemia.
5. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to:

   * Uncontrolled major seizure disorder
   * Unstable spinal cord compression
   * Any psychiatric disorder that prohibits obtaining informed consent.
   * Any other concurrent infectious disease requiring IV antibiotics within 2 weeks prior to the first dose of therapy
6. Patients with clinically significant cardiac disease including, but not limited to, any of the following

   * Myocardial infarction ≤ 6 months prior to first dose
   * Uncontrolled ventricular arrhythmia, recent (within 3 months)
   * Superior vena cava syndrome
   * Unstable angina pectoris
   * Uncontrolled congestive heart failure (New York Heart Association > class II)
   * Uncontrolled ≥ Grade 3 hypertension (per CTCAE)
   * Uncontrolled cardiac arrhythmias
7. Patients with a history of hemorrhagic or ischemic stroke within 6 months prior to enrollment
8. Patients with a history of cirrhotic liver disease (Child-Pugh Class B or C)
9. Persistent toxicities (>/= Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia or peripheral sensory neuropathy
10. Patients with duodenal stent or other GI disorder/defect that would interfere with absorption of oral medication

    o Includes patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
11. Patients with known untreated or symptomatic central nervous system (CNS) metastases
12. Prior known hypersensitivity reaction to study drugs and/or any of their excipients
13. Minor or major surgical procedure within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
14. Inability to comply with study and follow-up procedures
15. Patients deemed otherwise clinically unfit for clinical trial per investigators discretion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 50 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Determine the Safety of Combination Cirtuvivint with Olaparib | 6 months
  To determine the safety and tolerability of combination Cirtuvivint and Olaparib in BRCA/HRD platinum resistant ovarian cancer as evaluated by CTCAE v5.0 criteria.
Determine the recommended Phase 2 Dose of Cirtuvivint with Olaparib | 6 months
  To determine the recommended Phase 2 Dose (RP2D) and regimen of the combination therapy

SECONDARY OUTCOMES:
Evaluate the Cmax (peak plasma concentration) of Cirtuvivint when given in combination with olaparib | 3 years
  To evaluate the Cmax (peak plasma concentration) of Cirtuvivint when given in combination with olaparib
Evaluate the AUC (Area under the curve for plasma concentration) of Cirtuvivint when given in combination with olaparib | 3 years
  To evaluate the AUC (Area under the curve for plasma concentration) of Cirtuvivint when given in combination with olaparib
Evaluate the half-life (elimination half-life in plasma) of Cirtuvivint when given in combination with olaparib | 3 years
  To evaluate the half-life (elimination half-life in plasma) of Cirtuvivint when given in combination with olaparib
Evaluate CL (drug clearance) of Cirtuvivint when given in combination with olaparib | 3 years
  To evaluate CL (drug clearance) of Cirtuvivint when given in combination with olaparib

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Corr, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - CU Medicine Clinics, Aurora, Colorado
  - Universtiy of Colorado Hospital, Aurora, Colorado